CLINICAL TRIAL: NCT02528409
Title: A Double-Blind, Placebo-Controlled Study of Vortioxetine in the Treatment of Binge Eating Disorder
Brief Title: Vortioxetine for Binge Eating Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-1115
Record Dates: First submitted 2015-08-13; First posted 2015-08-19 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 10 milligrams per day for the first week and 10 milligrams per day for the final taper week 20 milligrams per day for 10 weeks between taper periods.
  Interventions: Drug: Placebo
- Vortioxetine (Experimental): 10 milligrams per day day for the first week and 10 milligrams per day for the final taper week 20 milligrams per day for 10 weeks between taper periods.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Medication currently approved for major depression.
  Other Names: Brintellix
  Arms: Vortioxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of the present study is to examine the efficacy and safety of vortioxetine vs placebo in adults with moderate to severe Binge eating disorder, as indicated by at least 3 binge eating days per week for the 2 weeks before the baseline visit.

DETAILED DESCRIPTION:
Binge-eating disorder recently included in the Diagnostic and Statistical Manual, 5th Edition, is now recognized as a serious public health problem. Binge-eating disorder is associated with obesity and psychiatric comorbidities, including depression, and may be predictive of metabolic syndrome. Many patients are undertreated despite functional impairments and personal and social difficulties leading to a poor quality of life. Binge-eating disorder is characterized by recurrent episodes of excessive food consumption accompanied by a sense of loss of control and psychological distress but without the inappropriate compensatory weight-loss behaviors of bulimia nervosa. Binge eating is seen in 23-46% of obese individuals seeking weight loss treatment and its severity relates to body mass index and predicts regain of lost weight.

Current treatments for binge eating disorder are often inadequate. Cognitive behavioral therapy has been shown to reduce binge eating but finding trained psychologists is difficult. Lisdexamfetamine was recently approved by the Food and Drug Administration for binge eating disorder but it carries risk of addiction and diversion and so will likely not be prescribed by most family physicians or psychiatrists. Other currently available medications, used off-label for binge eating disorder, include anticonvulsants, which may reduce binge eating but are often poorly tolerated. Therefore, additional clinical trials are needed to identify effective pharmacotherapies.

Consuming food is necessary for life and involves brain regions that are quite ancient in evolutionary terms. The intestinal tract itself is almost like a "second brain" in that it contains vast amounts of neurons used to transmit and process sensory information; indeed the intestinal tract contains more of the neurotransmitter serotonin than the brain itself. Peripheral signals from the body (including from the intestinal tract, but also from the blood stream - e.g. glucose levels) are transmitted to brain regions such as the hypothalamic nuclei to help regulate appetite/hunger and maintain equilibrium. Another key aspect of circuitry involved in eating involves the brain reward system, including the nucleus accumbens, which is regulated by neurotransmitters such as dopamine, opioids, noradrenaline, and serotonin. In humans, but to a lesser degree in other animals, there is also top-down control from the prefrontal cortices, which serve to regulate our behaviors and suppress our tendencies to crave rewards, and allow us to flexibly adapt our behavior rather than get stuck in repetitive habits. Thus, binge-eating most likely involves dysregulation of all three above domains regulating behavior: the primitive 'peripheral-hypothalamic' feedback system, reward circuitry, and top-down control circuitry. On a neurochemical level, binge eating may be related to dysfunction of the serotonergic, dopamine, glutamatergic, and norepinephrine systems. Thus, a medication to target binge eating needs to be multi-modal in terms of its pharmacology.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-65;
2. Primary diagnosis of Binge eating disorder;
3. At least 3 binge eating days per week for the 2 weeks before the baseline visit;
4. Ability to understand and sign the consent form.

Exclusion Criteria:

1. Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination (history of medical illness which is currently stable is allowed such as diabetes well controlled, treated hypothyroidism, hypertension, etc)
2. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
3. Subjects considered an immediate suicide risk based on the Columbia Suicide Severity rating Scale (C-SSRS) (www.cssrs.columbia.edu/docs)
4. Past 12-month DSM-5 major psychiatric disorder (psychotic disorder, bipolar disorder, major depressive disorder)
5. Past 6-month alcohol or substance use disorders
6. Illegal substance use based on urine toxicology screening
7. Initiation of psychological or weight-loss interventions within 3 months of screening
8. Use of any other prescription psychotropic medication (except an as needed hypnotic or as needed benzodiazepine)
9. Previous treatment with Vortioxetine
10. Currently taking over the counter weight loss medications. If willing to stop these medications, the participant will not be excluded based on this criterion.

10) Cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06; Primary Completion 2018-11 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Davis CA, Levitan RD, Reid C, Carter JC, Kaplan AS, Patte KA, King N, Curtis C, Kennedy JL. Dopamine for "wanting" and opioids for "liking": a comparison of obese adults with and without binge eating. Obesity (Silver Spring). 2009 Jun;17(6):1220-5. doi: 10.1038/oby.2009.52. Epub 2009 Mar 12. PMID 19282821
- [Background] Frisch MB, Cornell J, Villaneuva M (1993). Clinical validation of the Quality of Life Inventory: a measure of life satisfaction for use in treatment planning and outcome assessment. Psychol Assess 4:92-101.
- [Background] Gibb A, Deeks ED. Vortioxetine: first global approval. Drugs. 2014 Jan;74(1):135-45. doi: 10.1007/s40265-013-0161-9. PMID 24311349
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Hudson JI, Hiripi E, Pope HG Jr, Kessler RC. The prevalence and correlates of eating disorders in the National Comorbidity Survey Replication. Biol Psychiatry. 2007 Feb 1;61(3):348-58. doi: 10.1016/j.biopsych.2006.03.040. Epub 2006 Jul 3. PMID 16815322
- [Background] Johnson PM, Kenny PJ. Dopamine D2 receptors in addiction-like reward dysfunction and compulsive eating in obese rats. Nat Neurosci. 2010 May;13(5):635-41. doi: 10.1038/nn.2519. Epub 2010 Mar 28. PMID 20348917
- [Background] Kessler RC, Berglund PA, Chiu WT, Deitz AC, Hudson JI, Shahly V, Aguilar-Gaxiola S, Alonso J, Angermeyer MC, Benjet C, Bruffaerts R, de Girolamo G, de Graaf R, Maria Haro J, Kovess-Masfety V, O'Neill S, Posada-Villa J, Sasu C, Scott K, Viana MC, Xavier M. The prevalence and correlates of binge eating disorder in the World Health Organization World Mental Health Surveys. Biol Psychiatry. 2013 May 1;73(9):904-14. doi: 10.1016/j.biopsych.2012.11.020. Epub 2013 Jan 3. PMID 23290497
- [Background] Latagliata EC, Patrono E, Puglisi-Allegra S, Ventura R. Food seeking in spite of harmful consequences is under prefrontal cortical noradrenergic control. BMC Neurosci. 2010 Feb 8;11:15. doi: 10.1186/1471-2202-11-15. PMID 20141625
- [Background] Mahableshwarkar AR, Zajecka J, Jacobson W, Chen Y, Keefe RS. A Randomized, Placebo-Controlled, Active-Reference, Double-Blind, Flexible-Dose Study of the Efficacy of Vortioxetine on Cognitive Function in Major Depressive Disorder. Neuropsychopharmacology. 2015 Jul;40(8):2025-37. doi: 10.1038/npp.2015.52. Epub 2015 Feb 17. PMID 25687662
- [Background] Mathes WF, Brownley KA, Mo X, Bulik CM. The biology of binge eating. Appetite. 2009 Jun;52(3):545-553. doi: 10.1016/j.appet.2009.03.005. Epub 2009 Mar 20. PMID 19501749
- [Background] McElroy SL, Hudson JI, Capece JA, Beyers K, Fisher AC, Rosenthal NR; Topiramate Binge Eating Disorder Research Group. Topiramate for the treatment of binge eating disorder associated with obesity: a placebo-controlled study. Biol Psychiatry. 2007 May 1;61(9):1039-48. doi: 10.1016/j.biopsych.2006.08.008. Epub 2007 Jan 29. PMID 17258690
- [Background] McElroy SL, Guerdjikova AI, Mori N, O'Melia AM. Pharmacological management of binge eating disorder: current and emerging treatment options. Ther Clin Risk Manag. 2012;8:219-41. doi: 10.2147/TCRM.S25574. Epub 2012 May 8. PMID 22654518
- [Background] McElroy SL, Hudson JI, Mitchell JE, Wilfley D, Ferreira-Cornwell MC, Gao J, Wang J, Whitaker T, Jonas J, Gasior M. Efficacy and safety of lisdexamfetamine for treatment of adults with moderate to severe binge-eating disorder: a randomized clinical trial. JAMA Psychiatry. 2015 Mar;72(3):235-46. doi: 10.1001/jamapsychiatry.2014.2162. PMID 25587645
- [Background] Sheehan DV (1983). The Anxiety Disease. New York: Scribner's.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 10 milligrams per day for the first week and 10 milligrams per day for the final taper week 20 milligrams per day for 10 weeks between taper periods.
  Placebo
Period: Overall Study
Arm/Group | Placebo | Vortioxetine
Started | 40 | 40
Completed | 18 | 24
Not Completed | 22 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (12.9) | 41.4 (13.8) | 40.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 32 | 36 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 24 | 44
  White | 8 | 11 | 19
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Binge Eating Episodes
Description: Subjects will report the number of binge eating episodes in the week preceding the final visit (Week 12 of treatment), both to the investigator and via daily eating journals at all 9 visits. The outcome measure was the change in number of episodes from Week 0 (baseline) to the final visit (Week 12).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: binge eating episodes
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 28 | 29
binge eating episodes | .93 (1.49) | .76 (1.33)

2. Secondary Outcome: BMI
Description: Assessment of change in patient body mass index over the course of the study (from baseline to the final visit at Week 12).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 34 | 34
kg/m^2
  Pre-Treatment | 36.19 (8.47) | 38.39 (9.30)
  Post-Treatment | 36.29 (8.52) | 38.73 (9.66)

3. Secondary Outcome: Number of Participants With 4-week Cessation From Binge Eating
Description: Subjects will be assessed at 4 weeks to determine cessation of binge eating status.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 37 | 39
Participants
  No 4-Week Cessation | 27 | 26
  4-Week Cessation | 10 | 13

4. Secondary Outcome: Clinical Global Impression Improvement Scale (CGI)
Description: Patient global improvement relative to baseline, with scores ranging from 1-7. Higher scores indicate the patient is doing severely worse than they were at the beginning of treatment.
Time Frame: Week 12 (final) visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 33 | 33
units on a scale
  Pre-Treatment | 4.18 (.64) | 4.25 (.71)
  Post-Treatment | 2.79 (1.29) | 2.70 (1.33)

5. Secondary Outcome: Three-Factor Eating Questionnaire
Description: A self-reported measure of binge eating behavior that will be collected at all 9 study visits with scores ranging from 0-51, with higher scores indicating more compulsive eating habits.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 34 | 33
units on a scale
  Pre-Treatment | 7.71 (3.97) | 6.92 (4.53)
  Post-Treatment | 9.85 (5.12) | 9.48 (6.00)

6. Secondary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating
Description: A clinician-administered scale assessing binge eating severity that will be assessed at all 9 study visits. Scores range from 0-40 with higher scores indicating more severe OCD symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 34 | 33
units on a scale
  Pre-Treatment | 20.10 (4.03) | 20.55 (3.88)
  Post-Treatment | 10.44 (7.09) | 9.94 (8.10)

7. Secondary Outcome: Quality of Life Inventory
Description: A self-report assessment of patient perceived quality of life that will be assessed at baseline and final visit. The scale provides a discrete score ranging from -192 to 192, with higher numbers indicating higher subjective quality of life.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 18 | 21
units on a scale
  Pre-Treatment | 39.13 (29.00) | 35.00 (14.72)
  Post-Treatment | 46.22 (15.38) | 44.00 (16.69)

8. Secondary Outcome: Hamilton Depression Rating Scale
Description: A clinician-administered assessment of depression that will be assessed at all 8 study visits after the baseline visit. The scale provides a discrete score that ranges from 0-52, with higher scores indicating more severe depressive symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 34 | 34
units on a scale
  Pre-Treatment | 4.55 (4.32) | 4.32 (4.38)
  Post-Treatment | 2.06 (2.57) | 3.66 (4.38)

9. Secondary Outcome: Hamilton Anxiety Rating Scale
Description: A clinician-administered assessment of anxiety that will be assessed at all 9 study visits. The scale provides a discrete score that ranges from 0-56, with higher scores indicating more severe anxiety symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 33 | 32
units on a scale
  Pre-Treatment | 4.13 (4.26) | 3.68 (3.51)
  Post-Treatment | 1.79 (1.95) | 2.72 (4.18)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the 12 weeks of participation at every visit after the baseline visit (at each of the 8 follow-up visits -- each one or two weeks apart from each other, depending on the part of the study).
Arm/Group | Placebo | Vortioxetine
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 18/40 | 20/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Vortioxetine (N=40)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (9) | 10 (20)
Headache (Nervous system disorders) | 4 (5) | 4 (4)
Dizziness (Nervous system disorders) | 3 (5) | 4 (4)
Dry Mouth (Gastrointestinal disorders) | 2 (5) | 4 (5)
Insomnia (Nervous system disorders) | 2 (2) | 3 (7)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4)
Bloating (Gastrointestinal disorders) | 2 (3) | 3 (4)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Tingling/Numbness (Nervous system disorders) | 2 (2) | 1 (2)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Temperature Fluctuations (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (4)
Tooth Sensitivity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Panic symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
Blurry vision (Eye disorders) | 1 (1) | 1 (1)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (Nervous system disorders) | 1 (1) | 1 (1)
Loss of Libido (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Increased heart rate (Nervous system disorders) | 0 (0) | 1 (1)
Difficulty swallowing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Restlessness (Nervous system disorders) | 0 (0) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT02528409/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT02528409/ICF_001.pdf